CLINICAL TRIAL: NCT04080024
Title: A First-in-human Clinical Evaluation of the Novel Intravenous Contrast Agent SN132D in Patients With Breast and Pancreatic Cancer
Brief Title: A First-in-human Clinical Evaluation of SN132D in Patients With Breast and Pancreatic Cancer
Acronym: SPAGOPIX-01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Spago Nanomedical AB (Industry)
Collaborators: CTC Clinical Trial Consultants AB (Industry); Antaros Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SN132D CSP final version 6.0; 2018-002193-41 (EudraCT Number)
Record Dates: First submitted 2019-08-27; First posted 2019-09-06 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Breast Cancer; Pancreas Cancer
MeSH Terms: conditions — Breast Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single dose (i.v.) SN132D (Experimental)
  Interventions: Drug: SN132D

INTERVENTIONS:
Drug: SN132D — Novel manganese-based macromolecular MRI contrast agent

SUMMARY:
This phase I, first-in-human (FIH) study is open-label, non-randomised and non-placebo-controlled. The study is designed to evaluate the safety, tolerability and pharmacokinetics (PK) of a single intravenous dose of SN132D in approximately 24 patients with breast and pancreatic cancer. Magnetic resonance imaging (MRI) will be performed pre- and post-infusion of SN132D.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent including willingness to undertake 3 MRI investigations (30 minute each) in one day
2. Histological or cytological diagnosis of breast cancer > 5 mm (cT1c-cT4; cN0-cN3; Mx) or known or suspected pancreatic cancer with hepatic involvement with available or scheduled gadolinium enhanced MRI of the pancreas
3. At least 3 weeks between core needle biopsy and planned pre-dose MRI. Fine needle aspiration is allowed at any time before MRI.
4. Female and at least 18 years of age when signing the informed consent.
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1 at screening
6. Adequate renal and hepatic function: estimated glomerular filtration rate (eGFR) ≥ 50 mL/min/1.73 m2 (determined by the revised Lund-Malmö GFR estimating equation), bilirubin <1 x upper limit of normal (ULN; (in subjects with liver metastases <5 x ULN)), creatinine <1 x ULN, aspartate aminotransferase (ASAT) and alanine aminotransferase (ALAT) < 1 x ULN.

   Bilirubin ULN: 25 µmol/L, creatinine ULN: 90 µmol/L, ASAT ULN: 0.60 µkat/L and ALAT ULN: 0.75 µkat/L) at the screening visit.
7. Females of child-bearing potential* must agree to the use of effective contraception** or practice abstinence during the study and for 30 days after the IMP administration.
8. Adequate haematological function: haemoglobin ≥90 g/L, absolute neutrophil count (ANC) ≥1.3x109 /L and platelet count ≥ 100 x 109 /L.

   * A female of child-bearing potential is a sexually mature female who 1) has not undergone a hysterectomy or bilateral oophorectomy, or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e. had had menses at any time in the preceding 24 consecutive months).

     * Effective contraception is defined as contraceptive methods with a failure rate of < 1% to prevent pregnancy (combined [oestrogen and progestogen containing] hormonal contraception associated with inhibition of ovulation [oral, intravaginal, transdermal], progestogen-only hormonal contraception associated with inhibition of ovulation [oral, injectable, implantable], intrauterine device [IUD]or intrauterine hormone-releasing system [IUS]).

Exclusion Criteria:

1. Female patients who are pregnant or who are currently breast feeding.
2. Conditions contraindicating MRI including, but not limited to, body mass index (BMI) > 40 kg/m2 at screening claustrophobia, metallic implants or internal electrical devices (e.g., cochlear implant, nerve stimulator, gastric pacemaker, bladder stimulator, pacemaker, defibrillator, artificial valves in heart, aneurysm clips, etc.), and permanent makeup or tattoos which in the Investigator's opinion might jeopardise the patient's safety or interfere with the imaging measurements. The Investigator is encouraged to contact the MR clinic for advice on which implants, tattoos, etc may be unsuitable.
3. Other malignancy than breast and pancreatic cancer within the past 5 years with the exception of in situ removal of basal cell carcinoma or resected benign colonic polyps.
4. Moderate to severe hypertension as judged by the Investigator.
5. History of significant cardiovascular disease such as myocardial infarction, congestive heart failure, stroke, serious cardiac arrhythmias. History of angina within 6 months prior to screening.
6. Clinically diagnosed obstruction of bile duct as judged by investigator.
7. Prolonged QTcF (>450 ms), cardiac arrhythmias or any clinically significant abnormalities in the resting electrocardiogram (ECG) at the time of screening, as judged by the Investigator.
8. Abnormalities detected during examination at screening and admission, which in the opinion of the Investigator, may either put the patient at risk because of participation in the study or influence the results or the patient's ability to participate in the study.
9. Active infection requiring systemic treatment within one week prior to agent administration.
10. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the patient at risk because of participation in the study, or influence the results or the patient's ability to participate in the study.
11. Seropositive for human immunodeficiency virus (HIV), Hepatitis B surface antigen (HBsAg), or Hepatitis C virus (HCV) antibodies.
12. Any use of alcohol within 24 hours of admission to the clinic.
13. Plasma donation within 1 month of screening or any blood donation or corresponding blood loss during 3 months prior to screening.
14. Use of investigational agent within four weeks before Visit 1 or plans to initiate treatment with an investigational agent during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-08-23 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Number of treatment related adverse events (AEs) | Baseline up to 2 weeks
  Frequency, severity and seriousness of AEs including clinically significant changes in physical examinations, safety laboratory parameters, vital signs, electrocardiograms and injection site reactions will be assessed.

SECONDARY OUTCOMES:
Preliminary efficacy (MRI enhancing effect) | Day 1
  Preliminary efficacy will be evaluated by assessing changes between pre-dose images and post-dose images acquired using T1-weighted imaging sequences, analysing contrast-to-noise in primary tumour vs reference tissue, signal-to-noise in primary tumour, contrast-to-noise in liver and pancreas vs reference tissue and signal-to-noise in liver and pancreas. Additionally, Changes between pre-dose T1 and post-dose T1 in liver and pancreas will be analysed. In pancreatic cancer patients, presence or absence of liver metastases and a number of lesions and diameter of smallest and largest lesion in liver will also be analysed.
Pharmacokinetics as measured by area under the plasma concentration-time curve from time 0 to the last measurable time point (AUC0-t) for manganese (Mn) (mM x min) | Baseline up to Day 2
  Samples for pharmacokinetic analysis will be collected at predose and at 10 min, 20 min, 60 min, 65 min, 75 min, 90 min, 105 min, 3 h and 9 h post start of dosing.
Pharmacokinetics as measured by area under the plasma concentration-time curve from time 0 extrapolated to infinite time (AUCinf) for Mn (mM x min) | Baseline up to Day 2
  Samples for pharmacokinetic analysis will be collected at predose and at 10 min, 20 min, 60 min, 65 min, 75 min, 90 min, 105 min, 3 h and 9 h post start of dosing.
Pharmacokinetics as measured by maximum plasma concentration (Cmax) for Mn (µg Mn/mL) | Baseline up to Day 2
  Samples for pharmacokinetic analysis will be collected at predose and at 10 min, 20 min, 60 min, 65 min, 75 min, 90 min, 105 min, 3 h and 9 h post start of dosing.
Pharmacokinetics as measured by time to Cmax (Tmax) for Mn (h) | Baseline up to Day 2
  Samples for pharmacokinetic analysis will be collected at predose and at 10 min, 20 min, 60 min, 65 min, 75 min, 90 min, 105 min, 3 h and 9 h post start of dosing.
Pharmacokinetics as measured by plasma elimination half-life (T½) for Mn (h) | Baseline up to Day 2
  Samples for pharmacokinetic analysis will be collected at predose and at 10 min, 20 min, 60 min, 65 min, 75 min, 90 min, 105 min, 3 h and 9 h post start of dosing.
Pharmacokinetics as measured by total body clearance (CL) for Mn (L/h) | Baseline up to Day 2
  Samples for pharmacokinetic analysis will be collected at predose and at 10 min, 20 min, 60 min, 65 min, 75 min, 90 min, 105 min, 3 h and 9 h post start of dosing.
Pharmacokinetics as measured by apparent volume of distribution at steady state (Vss) for Mn (L) the terminal phase half-life (T½) for manganese (Mn) | Baseline up to Day 2
  Samples for pharmacokinetic analysis will be collected at predose and at 10 min, 20 min, 60 min, 65 min, 75 min, 90 min, 105 min, 3 h and 9 h post start of dosing.

OTHER OUTCOMES:
MRI enhancement of selected axillary (breast cancer patients) or regional and distant (e.g paraaortic lymph nodes, pancreatic cancer patients) lymph nodes | Day 1
  MRI enhancement of selected lymph nodes will be assessed by changes in contrast-to-noise vs reference tissue and signal-to-noise in selected lymph nodes between pre-dose images and 2 post-dose occasions
Visualization of the pancreatic duct | Day 1
  Visualization of the pancreatic duct will be assessed by a certified radiologist

CONTACTS AND LOCATIONS:
Overall Officials: Folke Sjöberg, MD, Prof, Principal Investigator — CTC Clinical Trial Consultants AB; Dan Curiac, MD, PhD, Principal Investigator — Gothia Forum Clinical Trial Center
Locations (2):
- Sweden (2):
  - Gothia Forum Clinical Trial Center, Gothenburg
  - CTC Clinical Trial Consultants AB, Uppsala

IPD SHARING:
Plan to Share IPD: No